CLINICAL TRIAL: NCT02133079
Title: Immunotherapy of Tumor With Autologous Tumor Derived Heat Shock Protein gp96
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cure&Sure Biotech Co., LTD (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-CIH-Li-01
Record Dates: First submitted 2014-05-03; First posted 2014-05-07 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Liver Cancer; Pancreatic Adenocarcinoma
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gp96 group (Experimental): autologous gp96 vaccination + basal treatment
  Interventions: Biological: autologous gp96 vaccination

INTERVENTIONS:
Biological: autologous gp96 vaccination — vaccination of autologous gp96 derived from tumor tissue + basal treatment

SUMMARY:
To evaluate the safety and effectiveness of autologous gp96 treatment of liver cancer and Pancreatic Adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and understand the informed consent document; must sign the informed consent;
2. Aged 18 to 75 years old , sex is not limited;
3. Pancreatic cancer or primary liver cancer,must have undergone radical resection;
4. Availability of at least 0.5 g tumor sample;
5. Receiving the first gp96 autologous immunotherapy within 8 weeks of postoperation;
6. Patients could not have received previous chemotherapy, radiation, or immunotherapy before 4 weeks of gp96 treatment；
7. ECOG ≤1；life expectancy of at least 12 weeks
8. Adequate bone marrow function including the absence of lymphopenia (ANC > 1,500/ mm3; Hemoglobin > 10g/dL ; platelet count >100,000/mm3), adequate liver function (serum glutamic oxaloacetic transaminase/ aspartate aminotransferase [AST], alanine amino transferase [ALT] <2.5 times institutional upper limit of normals [IULNs] and bilirubin (total) <1.5 times IULN), and adequate renal function (BUN and creatinine <1.5 times IULNs); 9. Agree to Surgical indications of Heart & lung and without the coagulation system disease;

10.Negative pregnancy test for female patients of childbearing potential; 11.Agree to use contraception or abstain from sexual activity from the time of consent through 3 month after the end of study drug administration.

Exclusion Criteria:

1. Unable to get the informed consent ;
2. Patient not suitable for radical resection;
3. Patients with active liver disease；
4. Did not get enough tumor tissue ;
5. Progression prior to vaccination as determined by the Principal Investigator;
6. Rreceiving other anti-cancer therapy at the same time;
7. Patient with allergic constitution;
8. Unstable or severe intercurrent medical conditions;
9. Current diagnosis of Human Immunodeficiency Virus and Patients with active uncontrolled infection;
10. Patients with any systemic disease needed to be treated with immunosuppressant or Corticosteroids;
11. Any other cilical trials within 30 days pre-vaccination;
12. Female patients who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2016-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
blood count | baseline
  blood count within 3 days before first vaccination
blood count | within 3 days after the second injection
  blood count within 3 days after the second injection
blood count | within 3 days after the 6th injection
  blood count within 3 days after the 6th injection
blood chemistries | baseline
  blood chemistries (including serum glutamic oxaloacetic transaminase/ aspartate aminotransferase [AST], serum alanine amino transferase [ALT], serum alkaline phosphatase, serum total bilirubin, serum blood urea nitrogen[BUN], serum creatinine, serum total protein and serum albumin) within 3 days before first vaccination
blood chemistries | within 3 days after the second injection
  blood chemistries (including serum glutamic oxaloacetic transaminase/ aspartate aminotransferase [AST], serum alanine amino transferase [ALT], serum alkaline phosphatase, serum total bilirubin, serum blood urea nitrogen[BUN], serum creatinine, serum total protein and serum albumin) within 3 days after the second injection
blood chemistries | within 3 days after the 6th injection
  blood chemistries (including serum glutamic oxaloacetic transaminase/ aspartate aminotransferase [AST], serum alanine amino transferase [ALT], serum alkaline phosphatase, serum total bilirubin, serum blood urea nitrogen[BUN], serum creatinine, serum total protein and serum albumin) within 3 days after the 6th injection
electrocardiogram | baseline
  electrocardiogram test within 3 days before first vaccination
electrocardiogram | within 3 days after the second injection
  electrocardiogram test within 3 days after the second injection
electrocardiogram | within 3 days after the 6th injection
  electrocardiogram test within 3 days after the 6th injection

SECONDARY OUTCOMES:
Disease-free survival | up to 3 years
overall survive | up to 3 years
changes in antigen specific T cells | baseline and within 3 days before the 6th injection
  tumor antigen specific T cells was determined by IFN-γ Enzyme-linked immunosorbent spot using the autologous tumor cell lysis as the antigen.

OTHER OUTCOMES:
Change from baseline in subpopulation of CD8+ T cells at the end of vaccination | within 3 days before the first vaccination, within 3 days after the 6th vaccination
  analysis of the expression of CCR7 & CD45RA of CD8+ T cells by FCM within 3 days before first vaccination and within 3 days after the 6th vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiang Cai, meidical, Principal Investigator — Cancer Insititute and Hospital,Chinese Academy of Medical Sciences; Lei Yu, medical, Principal Investigator — Cancer Insititute and Hospital,Chinese Academy of Medical Sciences
Locations (1):
- Cancer Insititute and Hospital,Chinese Academy of Medical Sciences, Beijing, China